CLINICAL TRIAL: NCT02256605
Title: Vitamin D3 Supplementation in Pediatric IBD: Weely vs Daily Dosing Regimens
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Collaborators: NASPGHAN Foundation (Other Government)
Responsible Party: Sponsor
Other Study IDs: 524835
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Inflammatory Bowel Disease (IBD)
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Insufficient Group: D-3 Chewable Wafer - 14,000 IU/wafer weekly Vitamin D-3 Caps - 2,000 IU/Cap daily Vitamin D-3 Liquid - 5,000 IU/ml (0.4) ml daily
  Interventions: Dietary Supplement: Vitamin D-3
- Deficient Group: D-3 Chewable Wafer - 50,000 IU/wafer weekly Vitamin D-3 Liquid - 5,000 IU/ml daily
  Interventions: Dietary Supplement: Vitamin D-3

INTERVENTIONS:
Dietary Supplement: Vitamin D-3 — Children with IBD, aged 5 to 17, who are vitamin D insufficient or deficient will be recruited at the time of a routine clinic visit or lab draw that included a 25(OH)D level as part of clinical practice/standard care. Once consent and assent are obtained, the children who are 25-hydroxyvitamin D [259OH)D] insufficient or deficient will be randomly assigned to a daily or weekly dosing regimen using block randomization to ensure equal group size.

SUMMARY:
The purpose of this prospecitve randomized controlled trial is to compare effectiveness and patient/family adherence of weekly or daily Vitamin D-3 dosing regimens in children with Inflammatory Bowel Disease (IBD) who are 25-hydroxyvitamin D [25(OH)D] insufficient or deficient. The primary aim of this pilot study is to evaluate the effectiveness of once weekly verses daily D-3 dosing regimens based on the most current IBD supplementation guidelines in improving 25(OH)D levels. A seconary aim is to determine if there is difference in adherence between dosing regimns.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 5 to 17 years with a diagnosis of Inflammatory Bowel Disease, who have a 25(OH)D level below 30 ng/ml within 2 weeks of enrollment
* Subject/family must be able and willing to take oral medications, complete a 3 day dietary record, and return for 8 week concluding visit or clinicl visit

Exclusion Criteria:

* Subjects will not be eligible if they are intolerant of vitamin supplementation or any ingredients in the chosen supplment, are unable or unwilling to take oral supplements, or are on specific medical therapy for diminished bone mineral density
* Children with parathryoid disease, granulomatous disorders or William's syndrome will also be excluded from the study

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with IBD, aged 5 to 17, who are vitamin D insufficient or deficient will be recruited at the time of a rountine clinic visit or lab draw that includes a 25(OH)D level as part of a clinical practice/standard of care.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
25 (OH)D level will be recorded at baseline and at 8 weeks as an absolute value (ratio data) and the percentage and direction (increase or decrease) of change between baseline and end of treatment level. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States